CLINICAL TRIAL: NCT05620043
Title: A Randomized, Single-center, Prospective Biopsy Study Comparing a Poly L-lactic Acid Biostimulator and a Calcium Hydroxylapatite Semi-permanent Filler
Brief Title: Gene Expression Study Between Two Dermal Injectables Hydroxylapatite Semi-permanent Filler
Acronym: Sculptra
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GLI.04.US.SL.020
Record Dates: First submitted 2022-11-07; First posted 2022-11-17 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2022-10

CONDITIONS: Gene Expression

STUDY DESIGN:
Intervention Model Description: Randomized, single-center, comparative study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Poly L-Lactic Acid (PLLA) (Active Comparator): Lyophilized PLLA with sodium carboxymethylcellulose, non-pyrogenic mannitol. Treatment needs to be reconstituted prior to injection, following product instruction.
  Interventions: Device: Sculptra
- Calcium Hydroxylapatite (CaHA) (Active Comparator): Opaque, sterile, non-pyrogenic, semi-solid, cohesive implant whose component is synthetic CaHA suspended in a gel carrier of glycerin, sodium carboxymethylcellulose, 0.3% lidocaine hydrochloride, and sterile water. Treatment injection follows product instruction.
  Interventions: Device: Radiesse Plus

INTERVENTIONS:
Device: Sculptra — Biostimulator
  Arms: Poly L-Lactic Acid (PLLA)
Device: Radiesse Plus — Semi-permanent filler
  Arms: Calcium Hydroxylapatite (CaHA)

SUMMARY:
To compare gene expression stimulated by a semi-permanent filler and a biostimulator via punch biopsy

DETAILED DESCRIPTION:
This is a randomized, single-center, comparative study to evaluate gene expression after treatment with a semi-permanent filler or a biostimulator.

This study is designed to enroll and randomize approximately 20 subjects in a 1:1 ratio of treatment to PLLA or CaHA. All randomized subjects are to have contour deficiency at the nasolabial folds.

Eligible subjects randomized to receive punch biopsy followed by treatment injection by the Treating Investigator at baseline. The method of injection was at the discretion of the Treating Investigator. A sufficient amount of product is injected to achieve optimal correction of the nasolabial folds, in the opinion of the Treating Investigator. PLLA group receives a second treatment at week 4 while CaHA group receives an optional touch-up if needed.

All subjects have final follow-up visit for a second punch biopsy on the other side of the nasolabial fold.

ELIGIBILITY:
Inclusion Criteria:

* Subject with a minimum of shallow nasolabial fold (NLF) contour deficiencies as assessed via the wrinkle assessment scale
* Subject with identical WAS scores on both NLFs
* Ability of giving consent for participation in the study
* Agreement to have skin biopsies on NLFs

Exclusion Criteria:

* Significant NLF asymmetry, or different WAS score on each NLF
* Pregnant, planning pregnancy during the course of the study or breastfeeding
* History of allergy or hypersensitivity to any ingredient of the treatment products
* History of allergy or hypersensitivity to anesthetics or lidocaine

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
Analyze gene expression via punch biopsy | 12 weeks after baseline
  Summary of fold change using by relative quantification method at week 12. Gene expression analysis is performed via qPCR processing using a panel of biomarkers related to scar tissue formation, collagen, elastin, extracellular matrix integrity, epidermal barrier, anti-aging, antioxidant, cell renewal/regeneration, inflammation, growth factor, and hydration among others.

SECONDARY OUTCOMES:
Evaluate volume change in the treated area using 3D imaging | 4 and 12 weeks after baseline
  Summary of total volume change in the nasolabial fold area measured by 3D photography at each visit. Total volume change corresponds to net volume change from baseline in the nasolabial fold.

CONTACTS AND LOCATIONS:
Overall Officials: Jill S Waibel, MD, Principal Investigator — Miami Dermatology & Laser Institute
Locations (1):
- Miami Dermatology & Laser Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Waibel J, Ziegler M, Nguyen TQ, Le JHTD, Qureshi A, Widgerow A, Meckfessel M. Comparative Bulk RNA-Seq Analysis of Poly-l-Lactic Acid Versus Calcium Hydroxylapatite Reveals a Novel, Adipocyte-Mediated Regenerative Mechanism of Action Unique to PLLA. Dermatol Surg. 2024 Nov 1;50(11S):S166-S171. doi: 10.1097/DSS.0000000000004425. PMID 39480040

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/43/NCT05620043/Prot_SAP_000.pdf